CLINICAL TRIAL: NCT07205692
Title: Multimorbidity and Cardiovascular Risk Factors After Renal Transplant
Acronym: MCaRT
Status: Recruiting | Type: Observational
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UHDB/2025/044
Record Dates: First submitted 2025-09-10; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Kidney Transplant; Cardiovascular (CV) Risk; Multimorbidity
Keywords: multimorbidity; kidney transplant; renal transplant; cardiovascular risk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Incident kidney transplants: Incident kidney transplants returning from surgical centre for follow up

SUMMARY:
Who can participate? Any adults over the age of 18 who have received a kidney transplant at the research centre are eligible for recruitment within the first month after transplant What does the study involve? The study involves observing and gathering data to understand how the health of people who receive a kidney transplant changes over the first year.

In particular the investigators are interested in the risk factors for heart disease and stroke, and how these change over the first year of transplant. The investigators are also interested in multiple health conditions, and how these impact patients after transplant.

There are no interventions but there will be measurements of diagnoses, risk factors for heart disease and stroke, and assessments of physical fitness Blood pressure, BMI, routine blood tests as well as assessing muscle and fat changes, how fit patients are and what new health conditions they have.

What are the possible benefits and risks of participating? There is no active treatment or intervention, so there are no risks of benefits compared to normal care.

Where is the study run from? University Hospitals of Derby and Burton NHS trust, at the Royal Derby hospital Renal Department.

When is the study starting and how long is it expected to run for? The study is expected to start 1/9/2025 and run for 2 years. Who is funding the study? The only costs of the study are funding for the staff member running the study, who is funded by the NIHR as an academic research fellow Who is the main contact? Dr Samuel Strain, Samuel.strain@nottingham.ac.uk

DETAILED DESCRIPTION:
1. BACKGROUND

   At the end of 2022 39,874 adult patients in the UK were living with a kidney transplant, representing 56.2% of the population on kidney replacement therapy. Kidney transplant remains the gold standard of renal replacement therapy and confers benefits in survival and quality of life over dialysis2. Short term survival post-transplant is good, with 94% adjusted 5 year survival in the UK for a transplant from a living donor and 87% for a deceased donor from the most recent UK renal registry data1.

   A high proportion of renal transplant patients have a high burden of comorbidities. Increasing multimorbidity has been shown in the general population to increase risk of premature death and hospital admissions and is associated with poorer function and greater economic costs. Much of the data in kidney transplant recipients focusses on comorbidity burden at time of transplant and the predictive use of this data for outcomes. There is little available data on the patterns and progression of multimorbidity for patients living with renal transplant. An assessment of the wider CKD cohort was undertaken using medical records and self reporting to understand multimorbidity, with a group of 176 transplant patients in the UK and showed that 92% had at least one comorbidity in addition to CKD. The most common comorbidity was hypertension (60.1%), followed by musculoskeletal conditions (40.9%) and then cardiovascular disease and diabetes. However, there is no data available, in this study or others, on the longitudinal development of comorbidities after transplant receipt. There is also no data available on the impact of multimorbidity on the quality of life of kidney transplant recipients. Although there is evidence for development of specific conditions, this has not been examined within the context of multiple long term health conditions.

   There is no consensus on the measurement of multimorbidity, and no consensus on which comorbid conditions should be used in a count. Expert reviewers suggest the conditions used to define multimorbidity should be guided by health impact and may be tailored to a study population. No such work has taken place in the kidney transplant population.

   A major comorbidity at time of transplantation and in post transplantation is cardiovascular disease and this is a major cause of death for patients with a renal transplant. Although the risk of adverse cardiovascular outcomes is decreased compared to patients on dialysis it is significantly increased compared to the general population. In addition, there is a high prevalence of both hypertension and diabetes within the transplant population. As well as these being common comorbidities to have at time transplant, patients commonly develop post-transplant diabetes. Alongside these factors, the risk of cardiovascular disease is also increased by raised BMI and lipid levels, which are commonly raised in renal transplant patients. The interaction between these risk factors and transplant specific factors such as immunosuppressive medication and post-transplant weight gain contribute to significant cardiovascular risk. There is no consensus on specific post-transplant treatment targets or interventions. Much of the evidence available for the timeline of development of cardiovascular risk factors is limited to retrospective cohort data and does not place cardiovascular disease within the context of multimorbidity6. In addition, much of the data predates current immunosuppression strategies and cardiovascular management strategies.

   Obesity is a significant factor in development of multimorbidity in the wider population7. In particular it is associated with development of cardiovascular risk factors and cardiovascular disease in the wider chronic kidney disease population as well as the transplant population. In the general population obesity contributes to frailty, and poor health-related quality of life, and can lead to worsening multimorbidity. There is also significant sarcopenia within the CKD and transplant population. Weight gain over the first year post transplant has been well recognised. However, assessing this using only body mass index (BMI) has limitations in the CKD and transplant populations as it does not take into account the possible normalisation of a pre-existing malnourished state. Using body composition techniques such as bio-impedance has shown changes in body composition post renal transplant, which has been related to muscle strength and fat distribution although this has not been correlated with function, multimorbidity, or development of cardiovascular risk factors.

   RATIONALE

   In this exploratory study the aim is to understand what happens to multimorbidity over the first year following transplant, including modifiable cardiovascular risk factors.

   The aim is to explore the development of multimorbidity on patients after kidney transplantation- the patterns of multimorbidity across conditions, common comorbidities, and progression of multimorbidity. The plan is to use a functional measure to understand how this might relate patient's experience.

   The study aims to measure the baseline characteristics of cardiovascular risk factors in the patient population as they return from transplant surgery to their referring centre, and then how these develop in the first year. The results of the study would aim to contribute to an evidence base regarding cardiovascular risk factors and identify targets for intervention within the first year. Early identification of modifiable risk factors can contribute to improvement of cardiovascular outcomes and graft survival.

   The study aims to use bioelectrical impedance to assess body composition and further understand the nature of weight gain post-transplant and how this relates to function, multimorbidity, exercise and other cardiovascular risk factors.

   The study aims also to recruit some patients into a qualitative study to help us understand possible barriers to improving modifiable cardiovascular risk factors with the aim of improving the effectiveness of any targeted interventions.

   Objectives

   Primary aims:

   • To assess the changes over time of multimorbidity in the one year post kidney transplantation

   Secondary aims:
   * To assess the changes over time of cardiac risk factors in the one year post kidney transplantation.
   * Understand the barriers to improved cardiovascular health and impact of multimorbidity using structured interviews.
   * Understand body composition changes over the one-year post transplant and how this relates to functional status Outcome

   STUDY DESIGN

   Study Part 1 The study is a prospective cohort study. Patients returning for follow up at the study centre post hospital discharge will be screened for eligibility. Demographic information will be recorded at baseline. This includes primary renal diagnosis, if participant had been on dialysis, type of dialysis and dialysis vintage. At each study visit the following data will be collected: eGFR (using the creatinine-based formula (CKD-EPI)), HbA1c, lipid levels, urine ACR, clinic blood pressure, weight, height, smoking status, functional status using the KDQOL 36 and sit to stand, comorbidities, medications. This will be done at the baseline visit, three months, 6 months and one year after initial study visit.

   Study Part 2 For those participating in the body composition element of the study this will take place at the baseline study visit, and at 6 months and one year after initial study visit. Patients must enter part 2 of the study at the first study visit. Patients must be entered into part 1 of the study to enter into part 2. All patients who enter the study will be offered part 2 of the study unless they are ineligible.

   Study Part 3 At the one-year study visit the investigators will recruit for the structured interview element of the study. This will take place as soon as can be arranged after this visit. The interviews will be carried out face to face. The aim is to recruit 10 participants for the interview. They will be recorded using trust recording equipment and transcribed and analysed by the research team. The plan is to use content analysis to understand the themes of barriers to healthy lifestyle and perceptions of health after renal transplantation. The plan is to screen and consent all participants until 10 are recruited for this element of the study.

   STUDY SETTING

   Study visits will be at the Royal Derby Hospital in the renal outpatient unit where participants attend for their usual renal outpatient appointments. Patients will be recruited from transplant coordinator data as they return from transplant.

   Recruitment

   Patient Identification

   Patients will be identified by the transplant coordinator on return to UHDB after transplant.

   All patients receiving a transplant will be screened and assessed by the eligibility criteria.

   Screening

   Once identified, the investigators will ask the potential participants if they were interested in the study, and a PIS will be provided at the time. Patients will be contacted either at a face-to-face clinic visit or via phone call for recruitment. The participants will be given time to read the PIS and at agreed time, recontacted to discuss any queries and check if they would like to consent for participation.

   Consent

   Informed consent must be obtained prior to the participant undergoing procedures that are specifically for the purposes of the study (including the collection of identifiable participant data, unless the study has prior approval from the Confidentiality Advisory Group (CAG) and the REC).

   Once potential participants have had sufficient time to consider the PIS and opportunity to discuss any questions, the investigator will take informed, written consent. Participants may withdraw consent at any point and will be withdrawn from the study.

   Translation services via the clinical setting (language line) will be available for those whom English is not their first language for all aspects of the study. Translation services for information sheets and consent forms will be available in other languages and also for study visits, phone calls and structured interviews if required.

   The Principal Investigator (PI) retains overall responsibility for the informed consent of participants at their site and must ensure that any person delegated responsibility to participate in the informed consent process is duly authorised, trained and competent according to the REC approved protocol and applicable guidelines and regulations.

   Study Assessments

   Data will be collected from medical records, confirmed with participants and entered into the CRF: Participants will have demographic information recorded at baseline. This will include age, primary renal diagnosis, dialysis modality and vintage, and transplant details including deceased or living donor, induction regime, and length of hospital stay for transplant operation.

   At each study visit collect the following data: eGFR (using the creatinine-based formula (CKD-EPI)), HbA1c, lipid levels, urine ACR, standardised office blood pressure, weight, height, smoking status, functional status, comorbidities, medications.

   Functional status will be assessed using the KDQOL SF 36 and a sit-to-stand test. This is a validated survey assessing quality of life for patients with kidney disease. KDQOL has been translated and validated in a number of languages and if these are available will be used when applicable, along-side translation services in place in the renal department when needed.

   For those in group 2 bioimpedance will be done at baseline, 6 months, and one year. Bioimpedance will involve the Inbody bioimpedance machine in the UHDB renal outpatients department.

   These involves participants wearing light clothing and takes approximately 5 minutes. This measures body composition, which divides weight into different components.

   The structured interview will take approximately 20 minutes, and will take place at the closest available outpatient clinic appointment to the one year follow up visit. This will be recorded via already available transcription devices and transcribed by the study team.

   Study visits will be aligned to the closest clinic appointment. Study visits will be at the first available opportunity after return to follow up at UHDB, then subsequently at one month, three months, six months and one year after this visit. Blood tests will be taken as part of usual standard of care and data collected from these results resulting in no extra blood tests for the patient.

   There will be no compensation for participants. The investigators will offer refreshments for the study assessments from within the department. If a patient requires transport this will be part of their normal clinic arrangements. The investigators discussed the format of the assessments with our local PPIE group who felt that the arrangements were satisfactory.

   Withdrawal Criteria

   Participants will be withdrawn from the study if they withdraw consent to participate at any time. Participants do not have to provide a reason for withdrawal of consent. Subjects will also be withdrawn if it is deemed unsafe or is found to be impossible to proceed in the opinion of the investigators.

   The participants will be made aware that this will not affect their future care. Participants will be made aware (via the information sheet and consent form) that should they withdraw the data collected to date cannot be erased and may still be used in the final analysis.

   Storage and Analysis of Samples

   No samples will be stored. Routine laboratory tests will be undertaken as per clinical practice in an NHS laboratory and samples destroyed after analysis. No additional research specific samples will be taken, the results from routine clinical tests will be used.

   End of Study

   The end of study will be defined as when the last 12 month follow-up visits are complete. The CI will notify the Sponsor, participating sites and REC within 90 days of the end of study. The clinical study report will be written within 12 months of the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Capable of giving informed consent
* In receipt of a single organ renal transplant and being followed up by UHDB as the referring team.

Exclusion Criteria:

• Graft failure before return to follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Incident kidney transplant recipients returning to referring centre
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Multimorbidity | One year after transplant
  The changes from baseline to year one of multimorbidity in the one year post kidney transplantation as measured by a disease count.

SECONDARY OUTCOMES:
Blood pressure | One year
  The changes over time at baseline, 3 months, 6 months and one year, within patients of blood pressure.
Lipid levels | One year
  The changes over time at baseline, 3 months, 6 months and one year, within patients of lipid levels
Weight | One year
  The changes over time at baseline, 3 months, 6 months and one year, within patients of weight
HbA1c | One year
  The changes over time at baseline, 3 months, 6 months and one year, within patients of HbA1c
Qualitative interview | One year after transplant
  Understand the barriers to improved cardiovascular health and impact of multimorbidity using structured interviews. This is a qualatative measure and will be completed using thematic analysis.
Skeletal muscle as assessed by bioimpedance in kg | One year after transplant
  Body composition analysis of measured skeletal muscle over the one-year post transplant from baseline to year one.
Body fat as measured by bioimpedance as percent body fat (the proportion of total body weight that is fat) | One year
  Change in body composition measured visceral body fat in one year after transplant- measured at baseline, 6 months and one year
Kidney Disease Quality of Life Instrument (KDQOL)- 36 | Over one year
  Changes in KDQOL-36 over the one year post transplant measured at baseline, 3 months, 6 months, and one year. Score from 0-100, higher scores indicate a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Selby, Principal Investigator — University of Nottingham and UHDB
Locations (1):
- Royal Derby Hospital, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2025-08-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT07205692/Prot_000.pdf